CLINICAL TRIAL: NCT01568541
Title: Fluoride Intake From Tooth Brushing With Children's and Regular Toothpastes: a Study With Preschooler Children
Brief Title: Fluoride Intake From Toothbrushig With Children's or Regular Toothpastes
Acronym: F
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: University of Campinas, Brazil (Other); State University of Montes Claros (Unknown); Coordination for the Improvement of Higher Education Personnel (Other); Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Principal Investigator, Carolina Castro Martins, Principal Investigator, Federal University of Minas Gerais
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: NCT17591320
Record Dates: First submitted 2012-03-28; First posted 2012-04-02 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Healthy Individuals
Keywords: children; dentifrice; fluoride; dental fluorosis
MeSH Terms: conditions — Fluorosis, Dental

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Children' toothpaste (Active Comparator): Children's toothpastes
  Interventions: Drug: Regular toothpastes
- Regular toothpastes (Active Comparator): Regular toothpastes
  Interventions: Drug: Children's toothpastes

INTERVENTIONS:
Drug: Regular toothpastes — One tooth brushing
  Arms: Children' toothpaste
Drug: Children's toothpastes — One tooth brushing
  Arms: Regular toothpastes

SUMMARY:
There are controversial data about fluoride intake by children when tooth brushing with children's or regular toothpastes. However, a study have showed that children were exposed to a dose of 0.051 mg F/Kg/day and 0.046 mg F/kg/day by tooth brushing with children's and and regular toothpaste, respectively. Fluorides doses were too close and is questioned if there is a real clinical relevance in terms of risk of dental fluorosis. It is important to evaluate if children's toothpastes does really represent a risk of fluoride intake when compared to the regular toothpastes in terms of risk of dental fluorosis. The hypothesis is that both children's and regular toothpastes can represente risks of development of dental fluorosis and can represent similar fluoride exposure by children.

DETAILED DESCRIPTION:
Subjects: Children at age of development of dental fluorosis (up to 4 years) enrolled at day care centres from the city of Montes Claros (0.7 ppm F), Brazil.

The study design has two phases:

1. In the first phase, children are required to bring at the day care centres the tooth brush and the toothpaste used at home. There is no randomization, since the inclusion in either children's or regular toothpaste groups will be done based on each child's preference. The children are requested to tooth brush as the usual manner that the parent and the child do at home. Saliva expectorates are collected as the protocol described by Guha-Chowdhury et al. (1996). No instructions are provided in this phase or interventions by the researcher. Saliva expectorates are collected for further laboratory analysis. Toothpastes are collected for laboratory analysis.
2. In the second phase, children are required to toothbrush with other type of toothbrush following the same tooth brushing protocol. For example, children that previously used children's toothpaste will be provided a regular toothpaste, and vice-versa.

Parents are requested to answer a questionnaire regarding their children's tooth brushing habits and socioeconomic factors.

Laboratory analysis provides estimation of fluoride intake from tooth brushing with both toothpastes.

Analysis will base on dose of fluoride intake (mg F/Kg body weight/day) considering children's and regular toothpastes.

ELIGIBILITY:
Inclusion Criteria:

1. Consent demonstrates understanding of the study and willingness to participate as evidenced by voluntary written of informed consent and has received a signed and dated copy of the informed consent form.
2. Age up to 48 months.
3. Compliance understands of the study and ability to comply with the study procedures.
4. Good oral health as considered by the investigator.
5. Good general health as considered by the investigator, with no clinically significant and/or relevant abnormalities of medical history.

Exclusion Criteria:

1. Children aging older than 48 months or younger of 6 months.
2. Parents who do not allow the child's participation.
3. Children that refuse to follow the study procedure.
4. Volunteers that do not complete the whole study protocol.

Ages: 6 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 208 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Evidence of mean dose of fluoride intake from tooth brushing with children's and regular toothpastes. | One week interval between two tooth brushings

SECONDARY OUTCOMES:
Fluoride concentrations in toothpastes used by children. | From date of toothpastes collection until laboratorial analysis, assessed up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Carolina C Martins, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (3):
- Brazil (3):
  - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - State University of Montes Claros, Montes Claros, Minas Gerais
  - Piracicaba School of Dentistry of State University of Campinas, Piracicaba, São Paulo

REFERENCES:
- [Background] Martins CC, Paiva SM, Lima-Arsati YB, Ramos-Jorge ML, Cury JA. Prospective study of the association between fluoride intake and dental fluorosis in permanent teeth. Caries Res. 2008;42(2):125-33. doi: 10.1159/000119520. Epub 2008 Mar 4. PMID 18319589
- [Background] Martins CC, Paiva SM, Cury JA. Effect of discontinuation of fluoride intake from water and toothpaste on urinary excretion in young children. Int J Environ Res Public Health. 2011 Jun;8(6):2132-41. doi: 10.3390/ijerph8062132. Epub 2011 Jun 10. PMID 21776221
- [Background] Oliveira MJ, Paiva SM, Martins LH, Ramos-Jorge ML, Lima YB, Cury JA. Fluoride intake by children at risk for the development of dental fluorosis: comparison of regular dentifrices and flavoured dentifrices for children. Caries Res. 2007;41(6):460-6. doi: 10.1159/000107933. Epub 2007 Sep 7. PMID 17823508
- [Result] Cury JA, Oliveira MJ, Martins CC, Tenuta LM, Paiva SM. Available fluoride in toothpastes used by Brazilian children. Braz Dent J. 2010;21(5):396-400. doi: 10.1590/s0103-64402010000500003. PMID 21180793
- [Result] Martins CC, Oliveira MJ, Pordeus IA, Cury JA, Paiva SM. Association between socioeconomic factors and the choice of dentifrice and fluoride intake by children. Int J Environ Res Public Health. 2011 Nov;8(11):4284-99. doi: 10.3390/ijerph8114284. Epub 2011 Nov 10. PMID 22163207